CLINICAL TRIAL: NCT03634501
Title: Clinical Study on Anti-tumor Effect Induced by Activated Primary Natural Killer（NK）Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Zhiguo Chen, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XuanWuH-NK
Record Dates: First submitted 2018-08-03; First posted 2018-08-16 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer; Breast Cancer; Colon Cancer; Pancreatic Cancer; Ovarian Cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells (Experimental): Activated NK from peripheral blood and/or umbilical cord blood（UCB）
  Interventions: Biological: Activated NK

INTERVENTIONS:
Biological: Activated NK — Cell suspension

SUMMARY:
This study will analyze and evaluate the following items:

1. The safety of natural killer（NK） cells for treatment of subjects with solid tumors. Forty patients will be enrolled for each of the five cancers (in total 200 patients will be enrolled).
2. The effectiveness of natural killer（NK）cell therapy alone or with chemotherapy or targeted drugs.

Subjects from 18 to 75 years of age who are diagnosed with a solid tumor including pancreatic cancer, lung cancer, breast cancer, ovarian cancer and colon cancer, and for whom standard treatments are not effective, may be eligible for this study. Participants undergo the following procedures:

Peripheral blood will be collected from a vein of arm. Peripheral blood mononuclear cells（PBMC） will be isolated and purified for NK manufacturing. After 14~21 days cultivation, activated NK will be harvested and formulated for clinical administration.

Subjects will receive NK cell treatment by intravenous infusion. The frequency is once every 3 or 4 weeks for the first 3 months. Participants who respond well after 3 months may be eligible to continue NK cell therapy; and those not may receive NK therapy combined with chemotherapy and/or targeted drugs, or chemotherapy/targeted drugs alone.

Evaluations during therapy including:

1. Clinical assessment, and history of medications;
2. Blood draws for routine and research tests, including but not limited to: lymphocyte population and circulating tumor cell analysis in peripheral blood;
3. CT scan, bone scan and positron emission tomography（PET ）scan, if indicated, for disease evaluation;
4. Pharmacokinetics study after NK infusion. For this test, the number of NK cells in the blood is measured over time at indicated time-points.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years (including boundary values);
2. Diagnosed with histologically and cellularly confirmed cancer of lung, breast, pancreas, ovary, or colon;
3. At least 8 weeks since any prior systemic therapy to treat the underlying malignancy (standard or investigational);
4. Life expectancy > 6 months, and performance status（KPS）> 60 points;
5. Organ functions meet the following criteria:

   1. Blood bilirubin < 2mg/dL,
   2. Aspartate transaminase（AST）<100 IU/L,
   3. Alanine transaminase（ALT） <100 IU/L,
   4. Creatinine <1.5 mg/dL,
   5. Urea nitrogen ≤ 25 mg/dL,
   6. Hemoglobin ≥ 9.0 g/dL,
   7. White blood cell count>3.5×109/L,
   8. Neutrophil count >1.5x109/L,
   9. Platelet count > 80 × 109 /L,
   10. Hematocrit >0.20,
6. No severe infections.

Exclusion Criteria:

1. Subjects who take combined systemic steroids within 2 weeks prior to treatment (except inhaled steroids);
2. Patients who take chemotherapy within 1 month prior to treatment;
3. Subjects receiving drugs that stimulate the production of bone marrow hematopoietic cells within two weeks prior to treatment;
4. Patients with T lymphoma and NK cell lymphoma;
5. Patients with autoimmune diseases, including but not limited to lupus erythematosus, rheumatoid arthritis, etc.;
6. Seriously uncontrollable infected patients;
7. Patients who are allergic to the biological agents in this treatment;
8. Patients with organ transplantation or organ failure;
9. Subjects with severe cardiovascular disease and severe renal failure;
10. Patients who are undergoing treatment of immunosuppressive drugs or long-term administration of immunosuppressive drugs after organ transplantation;
11. Patients with active infection or fever;
12. Subjects with severe cardiovascular and cerebrovascular diseases, diabetes and renal dysfunction;
13. Subjects with pregnancy or during the lactating period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity induced by NK infusion | 6 months
  The incidence of toxicity within each infusion within 6 months after NK administration

SECONDARY OUTCOMES:
Objective-response rate (ORR) | 6 months after 6 infusions of NK administration
  Objective-response rate (ORR): defined as the proportion of patients who achieve partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at any time on study.
Persistence of NK | Day 0, Day 7, Day30, Day 60, Day 90, Day 180
  Duration of NK persistence: defined as duration from Day 1 to the time when the NK level goes back to stable level

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Chen, PhD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided